CLINICAL TRIAL: NCT01646385
Title: Long-term Safety and Efficacy of Etanercept in a UK Observational Cohort Study - a Retrospective Database Analysis of British Society of Rheumatology Biologics Registry (BSRBR) Data
Brief Title: Study to Assess the Safety and Efficacy of Etanercept in Patients Treated Over the Long-term in Real-world Clinical Practice, Using Data Collected by the British Society of Rheumatology Biologics Registry
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801348
Record Dates: First submitted 2012-04-12; First posted 2012-07-20 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatoid Arthritis
Keywords: observational; non-interventional; cohort; retrospective; register; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- etanercept: adult rheumatoid arthritis patients initiating therapy with etanercept as their first biologic therapy
  Interventions: Drug: etanercept
- nbDMARD: biologic-naive adult rheumatoid arthritis patients with DAS28 >4.2 treated with non-biologic anti-rheumatic drugs(s).
  Interventions: Drug: non-biologic anti-rheumatic drugs

INTERVENTIONS:
Drug: etanercept — use as per routine clinical practice
  Groups: etanercept
Drug: non-biologic anti-rheumatic drugs — use as per routine clinical practice (methotrexate, azathioprine, cyclophosphamide, cyclosporine, leflunomide, other)
  Groups: nbDMARD

SUMMARY:
This study will assess the rates of serious adverse events and death in adult rheumatoid arthritis patients treated with etanercept over the long-term in real-life clinical practice. It will also assess whether there is any difference in the rate of serious adverse events in patients trated with etanercept in comparision to patients treated with conventional disease-modifying anti-rheumatic drugs (DMARDs). The study will in addition quantify the efficacy of etanercept in this population by assessing the rates of important clinical outcomes such as changes in disease activity and disability/functioning.

DETAILED DESCRIPTION:
patients recruited sequentially as seen in clinical practice

ELIGIBILITY:
Inclusion Criteria:

* adult
* rheumatoid arthritis
* group 1: initiating etanercept as first biologic therapy
* group 2: DAS28<4.2, biologic naive and treated with non-biologic DMARDs

Exclusion Criteria:

* diagnosis of other inflammatory arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with a diagnosis of rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 6393 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801348&StudyName=Study%20to%20assess%20the%20safety%20and%20efficacy%20of%20etanercept%20in%20patients%20treated%20over%20the%20long-term%20in%20real-world%20clinical%20practice%2C%20using%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Participants with active rheumatoid arthritis (RA) who received etanercept (ETN, as their first biological drug) in doses as per approved product label or summary of product characteristics (SmPC) were observed using the data in British Society for Rheumatology Biologics Register (BSRBR) for a maximum of 10 years. Doses of ETN and any concomitant medication could be adjusted according to medical and therapeutic necessity. Participants were eligible to receive any other therapy instead of ETN, as per investigator's discretion and the doses of these were not controlled in the follow-up.
- nbDMARDs: Biological naive participants with active RA who received non-biologic disease modifying anti-rheumatic drugs (nbDMARDs) in doses as per approved product label or SmPC were observed using the data in BSRBR for a maximum of 8.75 years. Doses of nbDMARDs and any concomitant medication could be adjusted according to medical and therapeutic necessity.
Period: Overall Study
Arm/Group | Etanercept | nbDMARDs
Started | 3529 | 2864
Completed | 2691 (Completed refers to participants who continued up to last follow-up.) | 1993 (Completed refers to participants who continued up to last follow-up.)
Not Completed | 838 | 871
Not completed — Death | 202 | 222
Not completed — Switched to alternate biologic | 636 | 649

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants treated with ETN or nbDMARDs who had a physician diagnosis of rheumatoid arthritis and a minimum of one consultant follow-up after baseline registration.
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept | nbDMARDs | Total
Number analyzed (Participants) | 3529 | 2864 | 6393
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (12.1) | 59.8 (12.4) | 57.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2727 | 2135 | 4862
  Male | 802 | 729 | 1531

OUTCOME MEASURES:

1. Primary Outcome: Crude Incidence Rate of Malignancy
Description: Participant-Year estimated by calculating all of the years that participants in a study were followed (number of evaluable participants multiplied by mean follow-up in years). Crude (unadjusted) incidence rate calculated as number of malignancy events divided by Participant-Year, multiplied by 1000.
Time Frame: Baseline up to last follow-up, assessed every 6 month for first 3 years and thereafter annually up to 10 years
Population: as for baseline characteristics
Measure: Number; unit: events per 1000 participant-years
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 3529 | 2864
events per 1000 participant-years | 14.7 | 23.9
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Cox proportional hazards model adjusted for age, baseline steroid, smoking history, previous cancer, and body mass index was used for analysis; Test type: Superiority or Other; p = 0.084, Regression, Cox; Hazard Ratio (HR) = 0.836, 95% CI 2-sided [0.683 to 1.025]

2. Primary Outcome: Crude Incidence Rate of Lymphoproliferative Malignancy (LM)
Description: Participant-Year estimated by calculating all of years that participants in a study were followed (number of evaluable participants multiplied by mean follow-up in years). Crude (unadjusted) incidence rate calculated as number of LMs divided by Participant-Year, multiplied by 1000. Lymphoproliferative: medical condition characterized by the dysfunction of the immune system often resulting in excessive production of lymphocytes. LMs included lymphoma, myeloma, and leukemia. Adverse outcome was defined as 'lymphoproliferative malignancy' in the field [lymphopro] labeled by BSRBR.
Time Frame: Baseline up to last follow-up, assessed every 6 month for first 3 years and thereafter annually up to 10 years
Population: as for baseline characteristics
Measure: Number; unit: events per 1000 participant-years
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 3529 | 2864
events per 1000 participant-years | 1.1 | 2.6
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Cox proportional hazards model adjusted for age was used for analysis; Test type: Superiority or Other; p = 0.035, Regression, Cox; Hazard Ratio (HR) = 0.512, 95% CI 2-sided [0.276 to 0.952]

3. Primary Outcome: Crude Incidence Rate of Serious Infections
Description: Participant-Year estimated by calculating all of the years that participants in a study were followed (number of evaluable participants multiplied by total follow-up in years). Crude (unadjusted) incidence rate calculated as number of serious infections divided by Participant-Year, multiplied by 1000. Serious infections included those infections which required intravenous antibiotics, hospitalization, or resulted in death. Adverse outcome was defined as 'serious infection' in the field [serinf] labeled by BSRBR.
Time Frame: Baseline up to last follow-up, assessed every 6 month for first 3 years and thereafter annually up to 10 years
Population: as for baseline characteristics
Measure: Number; unit: events per 1000 participant-years
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 3529 | 2864
events per 1000 participant-years | 35.1 | 36.2
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Cox proportional hazards model adjusted for age, gender, previous non-RA drugs, baseline steroid, baseline DMARDs, methotrexate, disease activity score based on 28-joints count (DAS28), and smoking history was used for analysis; Test type: Superiority or Other; p = 0.855, Regression, Cox; Hazard Ratio (HR) = 1.019, 95% CI 2-sided [0.831 to 1.251]

4. Primary Outcome: Crude Incidence Rate of Other Serious Adverse Events
Description: Participant-Year estimated by calculating all of the years that participants in a study were followed (number of evaluable participants multiplied by total follow-up in years). Crude (unadjusted) incidence rate calculated as number of other serious adverse events divided by Participant-Year, multiplied by 1000. Other serious adverse events were based on classifications assigned by the BSRBR and included cardiac serious adverse events (SAEs), central nervous system SAEs, and nonmalignant hematological SAEs.
Time Frame: Baseline up to last follow-up, assessed every 6 month for first 3 years and thereafter annually up to 10 years
Population: as for baseline characteristics
Measure: Number; unit: events per 1000 participant-years
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 3529 | 2864
events per 1000 participant-years | 20.3 | 29.6
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Cox proportional hazards model adjusted for age, gender, previous non-RA drugs, baseline steroid, methotrexate, and baseline health assessment questionnaire (HAQ) score was used for analysis; Test type: Superiority or Other; p = 0.001, Regression, Cox; Hazard Ratio (HR) = 0.700, 95% CI 2-sided [0.564 to 0.870]

5. Primary Outcome: Crude Incidence Rate of All-Cause Mortality
Description: Participant-Year estimated by calculating all of the years that participants in a study were followed (number of evaluable participants multiplied by total follow-up in years). Crude (unadjusted) incidence rate calculated as number of deaths divided by Participant-Year, multiplied by 1000. Death was recorded in the adverse outcomes table and in the consultant follow-up table. Where multiple events described death for the same participant, date of death was taken as per the earliest record.
Time Frame: Baseline up to last follow-up, assessed every 6 month for first 3 years and thereafter annually up to 10 years
Population: as for baseline characteristics
Measure: Number; unit: events per 1000 participant-years
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 3529 | 2864
events per 1000 participant-years | 12.0 | 20.1
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Cox proportional hazards model adjusted for age, gender, previous non-RA drugs, baseline steroid, methotrexate, baseline HAQ score, Charlson index, smoking history, and body mass index was used for analysis; Test type: Superiority or Other; p = 0.024, Regression, Cox; Hazard Ratio (HR) = 0.717, 95% CI 2-sided [0.537 to 0.958]

6. Secondary Outcome: Percentage of Participants Who Switched to Other Therapy Following Etanercept Discontinuation
Description: Participants who switched from etanercept to either DMARDs or alternative biologic drug are reported.
Time Frame: Baseline up to last follow-up, assessed every 6 month for first 3 years and thereafter annually up to 10 years
Population: Full Analysis set (FAS) population included all participants treated with ETN or nbDMARDs who had a physician diagnosis of rheumatoid arthritis and a minimum of one consultant follow-up after baseline registration. Only participants treated with ETN were to be analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 3529
percentage of participants
  Switched to DMARDs | 35.3
  Switched to alternative biologic | 18.0

7. Secondary Outcome: Time on Etanercept Therapy
Description: Time on etanercept therapy was calculated by Kaplan-Meier survival analysis.
Time Frame: Baseline up to last follow-up, assessed every 6 month for first 3 years and thereafter annually up to 10 years
Population: FAS population included all participants treated with ETN or nbDMARDs who had a physician diagnosis of rheumatoid arthritis and a minimum of one consultant follow-up after baseline registration. Only participants treated with ETN were to be analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Etanercept
Number analyzed (Participants) | 3529
years | 4.959 [4.539 to 5.379]

8. Secondary Outcome: Disease Activity Score Based on 28-Joints Count (DAS28) at Baseline
Description: DAS28 calculated from the number of swollen joints (SJC) and tender joints (TJC) using the 28 joints count, the serological markers of inflammation (erythrocyte sedimentation rate [ESR, millimeter per hour] or C-reactive protein [CRP, milligram per liter]) and patient's general health assessment (recorded on a Visual Analog Scale [VAS] of 0 millimeter [mm]-100 mm). DAS28 <=1.6 = remission, DAS28 <=2.4 = low disease activity, DAS28 >=3.2 to 5.1 = moderate disease activity, DAS28 >5.1 = severe disease activity.
Time Frame: Baseline
Population: FAS population included all participants treated with ETN or nbDMARDs who had a physician diagnosis of rheumatoid arthritis and a minimum of one consultant follow-up after baseline registration.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 3529 | 2864
units on a scale | 6.6 (1.0) | 5.6 (0.9)
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

9. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count (DAS28) at Year 1, 2, 3, 4, and 5
Description: DAS28 calculated from SJC and TJC using the 28 joints count, the serological markers of inflammation (ESR [millimeter per hour] or CRP [milligram per liter]) and patient's general health assessment (recorded on a VAS scale of 0 mm-100 mm). DAS28 <=1.6 = remission, DAS28 <=2.4 = low disease activity, DAS28 >=3.2 to 5.1 = moderate disease activity, DAS28 >5.1 = severe disease activity.
Time Frame: Baseline, Year 1, 2, 3, 4, 5
Population: FAS included all participants treated with ETN or nbDMARDs who had a physician diagnosis of rheumatoid arthritis and a minimum of 1 consultant follow-up after baseline registration. N (number of participants analyzed): participants evaluable for this measure, n: participants evaluable for specified time-points for each treatment arm, respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 3118 | 1356
units on a scale
  Change at Year 1 (n= 3118, 1356) | -2.16 [-2.21 to -2.11] | -1.42 [-1.51 to -1.33]
  Change at Year 2 (n= 2536, 1066) | -2.40 [-2.46 to -2.34] | -1.79 [-1.89 to -1.69]
  Change at Year 3 (n= 2141, 783) | -2.55 [-2.62 to -2.49] | -1.95 [-2.07 to -1.83]
  Change at Year 4 (n= 1623, 534) | -2.16 [-2.21 to -2.11] | -1.42 [-1.51 to -1.33]
  Change at Year 5 (n= 1351, 415) | -2.71 [-2.79 to -2.63] | -2.47 [-2.62 to -2.31]
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Change at Year 1: analysis was performed with Analysis of Covariance (ANCOVA) using the General Linear Model (GLM) method applying age, gender, baseline DAS28, previous non-RA drugs, baseline steroid, and baseline methotrexate as covariates; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Etanercept vs nbDMARDs; Change at Year 2: analysis was performed with ANCOVA using the GLM method applying age, gender, baseline DAS28, previous non-RA drugs, baseline steroid, and baseline methotrexate as covariates; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: Etanercept vs nbDMARDs; Change at Year 3: analysis was performed with ANCOVA using the GLM method applying age, gender, baseline DAS28, previous non-RA drugs, baseline steroid, and baseline methotrexate as covariates; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 4: Comparison: Etanercept vs nbDMARDs; Change at Year 4: analysis was performed with ANCOVA using the GLM method applying age, gender, baseline DAS28, previous non-RA drugs, baseline steroid, and baseline methotrexate as covariates; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 5: Comparison: Etanercept vs nbDMARDs; Change at Year 5: analysis was performed with ANCOVA using the GLM method applying age, gender, baseline DAS28, previous non-RA drugs, baseline steroid, and baseline methotrexate as covariates; Test type: Superiority or Other; p = 0.01, ANCOVA

10. Secondary Outcome: Percentage of Participants With Remission and Low Disease Activity as Assessed by Disease Activity Score Based on 28-Joints Count (DAS28)
Description: as for outcome 9
Time Frame: Year 1, 2, 3, 4, 5
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 3118 | 1356
percentage of participants
  Remission: Year 1 (n= 3118, 1356) | 13.0 | 12.6
  Remission: Year 2 (n= 2536, 1066) | 17.0 | 16.2
  Remission: Year 3 (n= 2141, 783) | 20.1 | 21.3
  Remission: Year 4 (n= 1623, 534) | 23.7 | 20.0
  Remission: Year 5 (n= 1351, 415) | 23.4 | 25.1
  Low disease activity: Year 1 (n= 3118, 1356) | 24.1 | 22.0
  Low disease activity: Year 2 (n= 2536, 1066) | 30.5 | 28.8
  Low disease activity: Year 3 (n= 2141, 783) | 34.1 | 33.2
  Low disease activity: Year 4 (n= 1623, 534) | 37.6 | 35.0
  Low disease activity: Year 5 (n= 1351, 415) | 37.3 | 43.4

11. Secondary Outcome: Time to Remission
Description: DAS28 calculated from SJC and TJC using the 28 joints count, the serological markers of inflammation (ESR [millimeter per hour] or CRP [milligram per liter]) and patient's general health assessment (recorded on a VAS scale of 0 mm-100 mm). DAS28 <=1.6 = remission, DAS28 <=2.4 = low disease activity, DAS28 >=3.2 to 5.1 = moderate disease activity, DAS28 >5.1 = severe disease activity. Time to achieve remission was calculated by Kaplan-Meier survival analysis.
Time Frame: Baseline up to last follow-up, assessed every 6 month for first 3 years and thereafter annually up to 10 years
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 3529 | 2864
years | NA [NA to NA] — Median time to remission could not be calculated as fewer than 50% of participants had achieved remission during the follow up period. | NA [NA to NA] — Median time to remission could not be calculated as fewer than 50% of participants had achieved remission during the follow up period.

12. Secondary Outcome: Health Assessment Questionnaire (HAQ) Score at Baseline
Description: HAQ: self-reported, valid assessment of functional disability in rheumatoid arthritis. Assessed based on ability of participants to perform daily activities in 8 categories: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. HAQ score range: 0-3: without any difficulty=0, with some difficulty=1, with much difficulty=2, unable to do=3. HAQ total scores expressed as overall mean score with range 0-3: 0-0.25=normal functioning; 0.25-0.5=mild functional limitation; 0.5-1=moderate functional limitation; more than 1=significant functional limitation.
Time Frame: Baseline
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 3529 | 2864
units on a scale | 2.1 (0.5) | 1.7 (0.7)
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

13. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score at Year 1, 2, and 3
Description: as for outcome 12
Time Frame: Baseline, Year 1, 2, 3
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 2291 | 1545
units on a scale
  Change at Year 1 (n= 2291, 1545) | -0.317 [-0.339 to -0.296] | -0.057 [-0.084 to -0.030]
  Change at Year 2 (n= 2071, 1203) | -0.309 [-0.333 to -0.286] | -0.062 [-0.095 to -0.030]
  Change at Year 3 (n= 1947, 995) | -0.301 [-0.326 to -0.277] | -0.064 [-0.100 to -0.027]
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Change at Year 1: analysis was performed with ANCOVA using the GLM method applying age, gender, baseline HAQ, previous non-RA drugs, baseline steroid, and baseline methotrexate as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Etanercept vs nbDMARDs; Change at Year 2: analysis was performed with ANCOVA using the GLM method applying age, gender, baseline HAQ, previous non-RA drugs, baseline steroid, and baseline methotrexate as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Etanercept vs nbDMARDs; Change at Year 3: analysis was performed with ANCOVA using the GLM method applying age, gender, baseline HAQ, previous non-RA drugs, baseline steroid, and baseline methotrexate as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA

14. Secondary Outcome: Percentage of Participants With Remission Based on Health Assessment Questionnaire (HAQ) Score
Description: HAQ: self-reported, valid assessment of functional disability in rheumatoid arthritis. Assessed based on ability of participants to perform daily activities in 8 categories: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. HAQ score range: 0-3: without any difficulty=0, with some difficulty=1, with much difficulty=2, unable to do=3. HAQ total scores expressed as overall mean score with range 0-3. Participants who had HAQ total score <=0.5 were considered in remission state.
Time Frame: Year 1, 2, 3
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 2291 | 1545
percentage of participants
  Year 1 (n = 2291, 1545) | 24.9 | 8.4
  Year 2 (n = 2071, 1203) | 23.6 | 8.0
  Year 3 (n = 1947, 995) | 23.9 | 7.2

15. Secondary Outcome: Health Assessment Questionnaire (HAQ) Score 6 Months Prior to And 6 Months Post-Switching Etanercept
Description: as for outcome 12
Time Frame: 6 months prior to and 6 months post switching etanercept
Population: FAS population. Here "N" (number of participants analyzed): participants evaluable for this measure, "n": participants evaluable for specified time-points. Only participants treated with ETN were to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 1227
units on a scale
  6-Months Prior to Switching (n = 1227) | 2.006 (0.625)
  6-Months Post-Switching (n = 754) | 2.017 (0.641)

ADVERSE EVENTS:
Description: Due to retrospective nature of the study, it was difficult to capture non serious adverse events (Non-SAEs) and only serious adverse events (SAEs) were captured.
Arm/Group | Etanercept | nbDMARDs
Serious Adverse Events (participants affected / at risk) | 944/3529 | 744/2864
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=3529) | nbDMARDs (N=2864)
Pneumonia (Infections and infestations) | 205 | 225
Septicaemia (Infections and infestations) | 34 | 28
Bone/Joint infection (Infections and infestations) | 83 | 31
Other serious infection (Infections and infestations) | 314 | 171
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 18
Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 7
Non-melanoma skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 79 | 79
Solid tumours (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 153 | 158
Congestive heart failure (Cardiac disorders) | 28 | 36
Myocardial infarction (Cardiac disorders) | 65 | 69
Other Cardiac events (Cardiac disorders) | 85 | 102
Central demyelination (Nervous system disorders) | 1 | 1
Optic neuritis (Nervous system disorders) | 2 | 0
Peripheral Neuropathy (Nervous system disorders) | 10 | 12
Other CNS event (Nervous system disorders) | 117 | 85
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopaenia (Blood and lymphatic system disorders) | 4 | 8
Agranulocytosis (Blood and lymphatic system disorders) | 2 | 0
Other dyscrasia (Blood and lymphatic system disorders) | 51 | 53
Leukopaenia (Blood and lymphatic system disorders) | 7 | 2
Pulmonary fibrosis (Blood and lymphatic system disorders) | 14 | 13
Death (General disorders) | 203 | 223
Lymphoproliferative (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.